CLINICAL TRIAL: NCT00244361
Title: A Phase I Clinical Trial of Rituximab for Pediatric Opsoclonus-Myoclonus Syndrome
Brief Title: Effectiveness of Rituximab in Pediatric OMS Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Pediatric Neuroinflammation Organization, Inc. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Michael R Pranzatelli, MD, National Pediatric Myoclonus Center/ SIU School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND #11,771; SCRIHS (04-112)
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Opsoclonus-myoclonus Syndrome; Opsoclonus; Myoclonus; Ataxia
Keywords: opsoclonus; myoclonus
MeSH Terms: conditions — Opsoclonus-Myoclonus Syndrome; Ocular Motility Disorders; Myoclonus; Ataxia | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rituximab

SUMMARY:
The purpose of this study is to reduce the symptoms of OMS by testing rituximab (Rituxan®), to remove B lymphocytes that make antibodies and trigger brain inflammation. Evidence suggests that autoimmune brain inflammation causes the symptoms of OMS. This study of blood and spinal fluid intends to find out what effect rituximab has on OMS and on the spinal fluid B-cells.

Rituximab targets and destroys B-cells, which make antibodies that can attack the brain and cause may OMS. It is infused through a vein over a period of several hours. Rituximab has been used widely and studied extensively since its approval in 1997 by the U.S. Food and Drug Administration (FDA) for non-Hodgkin's B-cell Lymphoma (NHL). Today, more than 300,000 patients have received rituximab, and it is part of more than 200 completed, ongoing, or planned clinical trials. Rituximab is not FDA-approved for OMS.

DETAILED DESCRIPTION:
Opsoclonus-myoclonus syndrome (OMS) is a rare but pervasive, paraneoplastic neurological disorder, purported to be autoantibody-mediated. We demonstrated expansion of B-cells in cerebrospinal fluid (CSF) despite tumor resection, chemotherapy, or conventional immunotherapy. Whether B-cells can be purged from the CSF compartment with benefit to the patient is unknown. Targeting of CSF B lymphocytes represents a novel and valuable paradigm shift in the therapy of centrally-mediated paraneoplastic disorders. The objective of this preliminary study is to determine if rituximab, a monoclonal antibody against CD20+ B-cells, reduces or eliminates CSF B-cells in OMS and whether the reduction results in clinical improvement. B lymphocyte subsets and relevant T-cell subsets will be immunophenotyped in the CSF and peripheral blood of children with OMS by four-color dual-laser flow cytometry. Sixteen children with an increased percentage of CSF B-cells will be treated with rituximab 375 mg/m2 IV once weekly for four consecutive weeks and CSF testing will be repeated at six months with more frequent clinical evaluations and blood testing out to 12 months. Clinical outcome will be rated blindly from videotapes by an experienced observer using a validated 12-item motor evaluation scale and quantifiable parameters of sleep, behavior and motor function. Immunological outcome variables will include percentages of B-cell subsets and quantitative immunoglobulins. Post-treatment results will be compared to pre-treatment values statistically. If rituximab proves to be an efficacious and safe method of treating CSF B-cell expansion and the neurological syndrome, this study will lead to a phase II trial with the eventual aim of gaining FDA approval of rituximab for this indication.

ELIGIBILITY:
Inclusion Criteria:

* written consent from parents
* have symptomatic OMS
* have CSF B-cell expansion (>1% B-cells)
* adequate renal function as indicated by normal BUN [10-25 mg/dL] and creatinine [0.4-1.2 mg/dL]
* adequate liver function, as indicated by up to 2x normal AST [0-35 U/L] and ALT [0-35 U/L].
* men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months after completion of treatment

Exclusion Criteria:

* treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (which ever is longer)
* receipt of a live vaccine within 4 weeks prior to enrollment
* previous treatment with Rituximab
* prior antibody therapy (does not include IVIg) within past 6 months
* history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* history of HIV (patients considered high risk will be screened)
* history of hepatitis B and/or hepatitis C (patients considered high risk will be screened)
* history of recurrent significant infection or history of recurrent bacterial infections
* known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment)
* significant cardiac (symptomatic arrhythmias or symptomatic structural heart disease) or pulmonary disease (including obstructive pulmonary disease)
* concomitant chemotherapy
* hemoglobin: >13.5 gm/dL or <10.0 gm/dL
* platelets: <100,000/mm or >500,000/mm K/cumm

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determine the effectiveness & selectivity of rituximab at depleting CSF B-cells in OMS with intrathecal B-cell expansion. This requires CSF & blood lympocyte immunophenotyping prior to the first infusion & intervals for 1 year after the final infusion.

SECONDARY OUTCOMES:
Evaluate the clinical efficacy & safety of rituximab by clinical assessments, scoring of videotapes for neurological severity, and various blood tests prior to the first infusion and then at one, three, six, and twelve months post the final infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Pranzatelli, M.D., Principal Investigator — National Pediatric Neuroinflammation Organization, Inc.
Locations (1):
- National Pediatric Myoclonus Center, Department of Neurology, SIU School of Medicine, 751 N Rutledge St, Springfield, Illinois, United States

REFERENCES:
- [Derived] Pranzatelli MR, Tate ED, Travelstead AL, Verhulst SJ. Chemokine/cytokine profiling after rituximab: reciprocal expression of BCA-1/CXCL13 and BAFF in childhood OMS. Cytokine. 2011 Mar;53(3):384-9. doi: 10.1016/j.cyto.2010.12.004. Epub 2011 Jan 5. PMID 21211990
- [Derived] Pranzatelli MR, Tate ED, Verhulst SJ, Bertolone SJ, Bhatla D, Granger M, Lebowizc J, Lockhart SK, Wiley JM. Pediatric dosing of rituximab revisited: serum concentrations in opsoclonus-myoclonus syndrome. J Pediatr Hematol Oncol. 2010 Jul;32(5):e167-72. doi: 10.1097/MPH.0b013e3181cf0726. PMID 20606544
- [Derived] Pranzatelli MR, Tate ED, Travelstead AL, Colliver JA. Long-term cerebrospinal fluid and blood lymphocyte dynamics after rituximab for pediatric opsoclonus-myoclonus. J Clin Immunol. 2010 Jan;30(1):106-13. doi: 10.1007/s10875-009-9335-3. Epub 2009 Oct 17. PMID 19838774